CLINICAL TRIAL: NCT02764268
Title: Apatinib Dose Titration: Analyses of Exposure, Safety and Efficacy in Advanced or Metastatic Gastric Cancer
Brief Title: Apatinib Dose Titration in Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: HR-APTN-DT-AGC
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2016-04

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Pharmacokinetics; Dose titration
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib (Experimental)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib

SUMMARY:
Apatinib dose titration in Advanced or Metastatic Gastric Cancer

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 70 years of age
2. Histological confirmed advanced or metastatic adenocarcinoma of the stomach
3. Have failed for at least 2 lines of chemotherapy
4. Life expectancy of at least 12 weeks
5. Eastern Cooperative Oncology Group Performance Status of 0 or 1
6. At least one measurable lesion beyond stomach (larger than 10 mm in diameter by spiral CT scan)
7. Duration from the last therapy is more than 6 weeks for nitroso or mitomycin
8. More than 4 weeks for operation or radiotherapy or cytotoxic agents
9. Adequate hepatic, renal, heart, and hematologic functions

Exclusion Criteria:

1. Pregnant or lactating women
2. History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
3. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)
4. Any factors that influence the usage of oral administration
5. Evidence of central nerves system metastasis
6. Intercurrence with one of the following: coronary artery disease, arrhythmia ,heart failure
7. proteinuria ≥ (+)
8. International Normalized Ratio > 1.5 and activated partial thromboplastin time > 1.5 × Upper limit of normal（ULN）
9. Certain possibility of gastric or intestine hemorrhage
10. Less than 4 weeks from the last clinical trial
11. Prior VEGFR inhibitor treatment
12. Disability of serious uncontrolled intercurrence infection Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, Pneumoconiosis, radiation pneumonitis, drug-related pneumonia, Pulmonary function damaged seriously etc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Interruptions | 15 months

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE(Common Terminology Criteria for Adverse Events) v4.0 | 15 months
Objective Response Rate(ORR) | 15 months
  Number of Participants Who Reached Complete Response and Partial Response Assessed by Recist(Response Evaluation Criteria in Solid Tumors)1.1 at the End of the Second Treatment Cycle.
Disease Control Rate(DCR) | 15 months
  Number of Participants Who Reached Complete Response and Partial Response and Stable Disease Assessed by Recist(Response Evaluation Criteria in Solid Tumors)1.1 at the End of the Second Treatment Cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Wang C, Zhang Y, Hao J, Yang N, Wang J, Peng M, Liu T, Zhang G, Zhan X, Zeng S, Zhang Y, Gao Y, Yao Y. Multiple-dose up-titration study to evaluate the pharmacokinetics, safety and antitumor activity of apatinib in advanced gastric adenocarcinoma. Front Oncol. 2022 Oct 18;12:876899. doi: 10.3389/fonc.2022.876899. eCollection 2022. PMID 36330490